CLINICAL TRIAL: NCT05183035
Title: A Randomized Phase 3 Trial of Fludarabine/Cytarabine/Gemtuzumab Ozogamicin With or Without Venetoclax in Children With Relapsed AML
Brief Title: Venetoclax in Children With Relapsed Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PedAL BCU, LLC (Other)
Collaborators: Princess Maxima Center for Pediatric Oncology (European Sponsor) (Unknown); AbbVie (Industry); Roche-Genentech (Industry); EuPAL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCC-101/APAL2020D; 2021-003212-11 (EudraCT Number); 2023-510160-12-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Venetoclax; Gemtuzumab Ozogamicin; Fludarabine; Cytarabine; Relapsed refractory; Azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cytarabine; Gemtuzumab; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Control Arm without Venetoclax (Active Comparator): During Cycle 1 (42-day-cycles), participants will receive 30 mg/m^2 of fludarabine followed by 2 g/m^2 of cytarabine on Days 1-5. Gemtuzumab 3 mg/m^2 will be given on Day 6 (only for participants with CD33 expression on leukemia blasts).
  During Cycle 2 participants will receive 30 mg/m^2 of fludarabine followed by 2 g/m^2 of cytarabine on Days 1-5. After Cycle 2 participants are assessed for HSCT or azacitidine maintenance therapy.
  Interventions: Drug: Fludarabine; Drug: Cytarabine; Drug: Gemtuzumab Ozogamicin; Drug: Azacitidine
- Arm B: Experimental Arm with Venetoclax (Experimental): During Cycle 1 (42-day-cycles), participants will receive 300 mg adult dose equivalent of venetoclax once on Day 1 followed by 600 mg adult dose equivalent of venetoclax on Days 2-21. Participants will also receive 30 mg/m^2 of fludarabine followed by 2 g/m^2 of cytarabine on Days 8-12. Gemtuzumab 3 mg/m^2 will be given on Day 13 (only for participants with CD33 expression on leukemia blasts).
  During Cycle 2, participants will receive 600 mg adult dose equivalent of venetoclax on Days 1-21. Participants will receive 30 mg/m^2 of fludarabine followed by 2 g/m^2 of cytarabine on Days 1-5. After Cycle 2 participants are assessed for HSCT or azacitidine maintenance therapy in combination with venetoclax.
  Interventions: Drug: Fludarabine; Drug: Cytarabine; Drug: Gemtuzumab Ozogamicin; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Fludarabine — Intravenous (IV) infusion
Drug: Cytarabine — Intravenous (IV) infusion
Drug: Gemtuzumab Ozogamicin — Intravenous (IV) infusion
Drug: Azacitidine — Intravenous (IV) infusion or subcutaneous injection
Drug: Venetoclax — Orally via tablet or powder suspension
  Arms: Arm B: Experimental Arm with Venetoclax

SUMMARY:
A study to evaluate if the randomized addition of venetoclax to a chemotherapy backbone (fludarabine/cytarabine/gemtuzumab ozogamicin [GO]) improves survival of children/adolescents/young adults with acute myeloid leukemia (AML) in 1st relapse who are unable to receive additional anthracyclines, or in 2nd relapse.

DETAILED DESCRIPTION:
Relapse of AML is driven by chemotherapy resistant stem cells. One mechanism of chemotherapeutic resistance in AML is the overexpression of the protein B-cell lymphoma 2 (BCL-2), an anti-apoptotic protein which sequesters intracellular activators of apoptosis. Venetoclax is a selective, potent, orally bioavailable, small molecule inhibitor of BCL-2 that restores programmed cell death in cancer cells.

This is a trial for children, adolescents and young adults with 2nd relapsed AML or 1st relapsed AML unable to receive additional anthracycline.

This is randomized trial of venetoclax in combination with intensive chemotherapy (fludarabine/cytarabine/gemtuzumab ozogamicin) for the first two cycles (42-day-cycles) that would inform and evaluate if this agent is an effective option for this population to improve its poor prognosis. Participants can receive up to two cycles of induction chemotherapy before hematopoietic stem cell transplantation (HSCT). If participants who have perceived clinical benefit cannot be transplanted after the 2 cycles, maintenance treatment may be given at the discretion of the investigator. In Arm B (experimental arm), participants can continue venetoclax if they have perceived clinical benefit, and maintenance therapy will combine venetoclax with azacitidine for a maximum of 24 cycles. In Arm A (control arm), participants will receive azacitidine in monotherapy. Maintenance is continued until clinical progression or unacceptable toxicity with a maximum of 24 cycles.

ELIGIBILITY:
Inclusion Criteria

* Participants must have enrolled on APAL2020SC, NCT Number: NCT04726241 prior to enrollment on ITCC-101/APAL2020D. (This is only applicable for participants in USA/Canada/Australia/New Zealand sites/Blood Cancer United territory).
* Participants must be ≥ 29 days of age and ≤ 21 years of age at enrollment.
* Participants must have one of the following:

  1. Children, adolescents, and young adults with AML without demonstrated FLT3/internal tandem duplication (ITD) mutation. Ideally, the status of the mutation needs to be proven in the current relapse. Nevertheless, patients with previous FLT3/ITD negative test from prior lines can be included based on local results in order to not delay the start of treatment.
  2. And participants must have AML which is either:

     * Untreated second relapse, in participants who are sufficiently fit to undergo another round of intensive chemotherapy, or
     * Untreated first relapse, in participants who cannot tolerate additional anthracycline containing chemotherapy per investigator discretion.
* Participants must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2 (≥ 50% Lansky or Karnofsky score).
* Participants must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to start of protocol treatment:

  1. Cytotoxic chemotherapy: Must not have received cytotoxic chemotherapy within 14 days prior to start of protocol treatment, except for corticosteroids, low dose cytarabine or hydroxyurea that can be given up to 24 hours prior to start of protocol treatment.
  2. Intrathecal cytotoxic therapy: No wash-out time is required for participants having received any combination of intrathecal cytarabine, methotrexate, and/or hydrocortisone.
  3. Antibodies: ≥ 21 days must have elapsed from infusion of last dose of an antibody-drug conjugate before start of protocol treatment. For unmodified antibodies or T cell engaging antibodies, 2 half-lives must have elapsed before start of protocol treatment. Any toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.
  4. Interleukins, Interferons and Cytokines (other than Hematopoietic Growth Factors): ≥ 21 days after the completion of interleukins, interferon or cytokines (other than Hematopoietic Growth Factors) before start of protocol treatment.
  5. Hematopoietic growth factors: ≥ 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or ≥7 days for short-acting growth factor before start of protocol treatment.
  6. Radiation therapy (RT) (before start of protocol treatment):

     * ≥ 14 days have elapsed for local palliative RT (small port);
     * ≥ 84 days must have elapsed if prior craniospinal RT or if ≥ 50% radiation of pelvis;
     * ≥ 42 days must have elapsed if other substantial bone marrow (BM) radiation.
  7. Stem Cell Infusions (before start of protocol treatment):

     * ≥ 84 days since allogeneic (non-autologous) bone marrow or stem cell transplant (with or without total body irradiation [TBI]) or boost infusion (any stem cell product; not including donor lymphocyte infusion [DLI]);
     * No evidence of active graft versus host disease (GVHD).
  8. Participants who are receiving cyclosporine, tacrolimus or other agents to treat or prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial. Participants must be off medications to treat or prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant for at least 14 days prior to enrollment.
  9. Cellular Therapy: ≥ 42 days after the completion of donor lymphocyte infusion (DLI) or any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.) before start of protocol treatment.
  10. Participants with prior exposure to venetoclax are eligible in this trial.
* Adequate organ function:

  1. Adequate Renal Function defined as:

     * Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 60ml/min/1.73 m^2, or
     * Normal serum creatinine based on age/sex
  2. Adequate Liver Function defined as:

     * Direct bilirubin < 1.5 x upper limit of normal (ULN), and
     * Alkaline phosphatase ≤ 2.5 x ULN, and
     * Serum glutamic pyruvic transaminase (SGPT) alanine aminotransferase (ALT) ≤ 2.5 x ULN. If higher transaminases outside these ranges (up to 5x ULN) are due to a radiographically identifiable leukemia infiltrate, the participant will remain eligible. Transaminase elevation up to 5x ULN is also allowed in case of steatosis on echography.
  3. Cardiac performance: Minimum cardiac function defined as:

     * No history of congestive heart failure in need of medical treatment
     * No pre-treatment diminished left ventricular function on echocardiography (shortening fraction [SF] < 25% or ejection fraction [EF] < 40%)
     * No signs of congestive heart failure at presentation of relapse.
* Participant, parent or guardian must sign and date informed consent and pediatric assent (when required), prior to the initiation of screening or study specific procedures, according to local law and legislation.

Exclusion Criteria

* Participants who in the opinion of the investigator may not be able to comply with the study requirements of the study, are not eligible.
* Participants with Down syndrome.
* Participants with Acute promyelocytic leukemia (APL) or Juvenile myelomonocytic leukemia (JMML).
* Participants with isolated CNS3 disease or symptomatic CNS3 disease.
* Participants with malabsorption syndrome or any other condition that precludes enteral administration of venetoclax.
* Participants who are currently receiving an investigational drug other than those specified for this study.
* Participants with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known congenital bone marrow failure syndrome.
* Participants with known prior allergy to any of the medications used in protocol therapy.
* Participants with documented active, uncontrolled infection at the time of study entry.
* Known hepatitis C virus (HCV), hepatitis B virus (HBV) (known positive hepatitis B virus (HBV) surface antigen (HBsAg) results), or human immunodeficiency virus (HIV) infection.
* Concomitant Medications

  * Participants who have received strong and moderate CYP3A inducers such as rifampin, carbamazepine, phenytoin, and St. John's wort within 7 days of the start of study treatment.
  * Participants who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit within 3 days of the start of study treatment.
  * Participants who have hypersensitivity to the active substance or to any of the excipients listed in summary of product characteristics (SPC).
* Pregnancy or Breast-Feeding:

  * Participants who are pregnant or breast-feeding.
  * Participants of reproductive potential may not participate unless they have agreed to use a highly effective contraceptive method per Clinical Trial Facilitation Group (CTFG) guidelines for the duration of study therapy and at least 30 days after last dose of venetoclax, or 7 months after gemtuzumab ozogamicin treatment, or for 6 months after the completion of all study therapy, whichever is longer.
  * Male participants must use a condom during intercourse and agree not to father a child or donate sperm during therapy and for the duration of study therapy and at least 30 days after last dose of venetoclax or 4 months after last dose of gemtuzumab ozogamicin, 6 months from the last dose of cytarabine, or 90-days after last exposure to any other chemotherapy, whichever is longer.

Additional criteria to receive a gemtuzumab ozogamicin infusion:

Gemtuzumab ozogamicin should not be given:

* to participants with history of veno-occlusive disease (VOD)/Sinusoidal obstruction syndrome (SOS) grade 3 or 4
* to participants with CD33 negative leukemic blasts (determined at local lab)

Note that these participants are eligible for the study but will not be treated with gemtuzumab ozogamicin.

Ages: 29 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 5 years

SECONDARY OUTCOMES:
Morphology Event Free Survival (EFS) | Up to 5 years
Flow-based Event Free Survival (EFS) | Up to 5 years
Flow-based Overall Response Rate (ORR) | Up to Day 84
Morphological Overall Response Rate (ORR) | Up to Day 84
Duration of Response (DOR) | Up to 5 years
Cumulative Incidence of Relapse (CIR) | Up to 5 years
Disease-related Mortality | Up to 5 years
Non-disease-related Mortality | Up to 5 years
Hematopoietic Stem Cell Transplantation (HSCT) Rate | Up to 5 years
Number of Participants with Adverse Events (AEs) | Up to 5 years
Maximum Observed Plasma Concentration (Cmax) of Venetoclax | Pre-dose, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 8 and Day 13 (cycle is 42 days); once on follow-up visits of Cycle 2 between Day 5 and Day 21
Time to Maximum Observed Plasma Concentration (Tmax) of Venetoclax | Pre-dose, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 8 and Day 13 (cycle is 42 days); once on follow-up visits of Cycle 2 between Day 5 and Day 21
Area Under the Plasma Concentration-time Curve Over a 24-hour Dose Interval (AUC0-24) | Pre-dose, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 8 and Day 13 (cycle is 42 days); once on follow-up visits of Cycle 2 between Day 5 and Day 21
Number of Participants That Are Pediatric Minimal Residual Disease (Ped-MRD) Negative with Complete Remission (CR), Partial Complete Remission (CRp), or Complete Remission with Incomplete Hematologic Recovery (CRi) | Up to 5 years
Number of Participants with International Working Group Complete Response (IWG-CR) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seth Karol, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (89):
- United States (44):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - MemorialCare Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital of Orange County Main Campus - Orange, Orange, California
  - Benioff Children's Hospital - Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Shands Children's Hospital, Gainesville, Florida
  - Nemours Children's Specialty Care Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital - Orlando, Orlando, Florida
  - Saint Joseph's Hospital - Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital - Adele Hall Campus, Kansas City, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Alliance for Childhood Diseases dba Cure 4 The Kids Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center, HMH, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center - New York, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - The Royal Children's Hospital - Children's Cancer Centre, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Sankt Anna-Kinderspital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen, Belgium
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Izaak Walton Killam (IWK) Health Center, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - SickKids - The Hospital for Sick Children, Toronto, Ontario
- Fakultni nemocnice v Motole, Prague, Prague, Czechia
- Rigshospitalet, Copenhagen, Capital Region, Denmark
- Uusi Lastensairaala, Helsinki, Etelä-Suomen Lääni, Finland
- France (6):
  - CHU de Toulouse - Hôpital des Enfants, Toulouse, Haute-Garonne
  - Hôpital Jeanne de Flandre, Loos, Hauts-de-France
  - CHU de Nantes - Hôpital Femme-Enfant-Adolescent, Nantes, Loire-Atlantique
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon, Rhône
  - Hôpital Armand-Trousseau, Paris, Île-de-France Region
  - Hôpital Universitaire Robert-Debré, Paris, Île-de-France Region
- Germany (5):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Padiatrische Hamatologie und Onkologie, Münster
  - Universitätsklinikum Münster, Münster
- Schneider Children's Medical Center of Israel, Petach Tikvah, Central District, Israel
- Italy (4):
  - Istituto Giannina Gaslini, Genova, Genoa
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza and Brianza
  - Ospedale Pediatrico Bambino Gesù, Roma, Rome
  - Ospedale Infantile Regina Margherita, Torino, Turin
- Japan (5):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya, Aiti
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Saitama Prefectural Children's Medical Center, Saitama-Shi, Saitama
  - National Center for Child Health and Development, Setagaya-Ku, Tokyo
  - Osaka City General Hospital, Osaka
- Prinses Maxima Centrum Kinderoncologie, Utrecht, Netherlands
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- Oslo Universitetssykehus, Oslo, Norway
- Instituto Portugues De Oncologia De Lisboa Francisco Gentil, Lisbon, Lisbon District, Portugal
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario La Fe, Valencia
- Karolinska Universitetssjukhuset Solna, Stockholm, Stockholm County, Sweden
- Universitaets - Kinderspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badawi M, Gopalakrishnan S, Engelhardt B, Palenski T, Karol SE, Rubnitz JE, Menon R, Salem AH. Dosing of Venetoclax in Pediatric Patients with Relapsed Acute Myeloid Leukemia: Analysis of Developmental Pharmacokinetics and Exposure-Response Relationships. Clin Ther. 2024 Oct;46(10):759-767. doi: 10.1016/j.clinthera.2024.09.008. Epub 2024 Oct 5. PMID 39368878